CLINICAL TRIAL: NCT01248702
Title: A Critical Pathway for Implantable Cardioverter-Defibrillators in Patients With Ischemic Cardiomyopathy
Acronym: CAPTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H10-01537
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Myocardial Infarction; Heart Failure
Keywords: Myocardial Infarction; Heart Failure; Sudden Cardiac Death; Critical Pathways
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Critical Pathway (Experimental)
  Interventions: Other: Use of the ICD Critical Pathway
- Standard Practice (No Intervention)

INTERVENTIONS:
Other: Use of the ICD Critical Pathway — The critical pathway is a series of predetermined processes designed to assess a patient's eligibility for an ICD. The critical pathway will incorporate current evidence-based practice guidelines.
  Other Names: ICD Critical Pathway
  Arms: Critical Pathway

SUMMARY:
The purpose of this study is to develop and implement a critical pathway to identify patients with ischemic cardiomyopathy who are candidates for an implantable cardioverter-defibrillator (ICD). This study will also determine whether the use of the critical pathway for ICDs is associated with a change in the ICD referral and implantation rate.

DETAILED DESCRIPTION:
Despite improvements in both medical management and revascularization strategies, sudden death is still a significant complication in patients with ischemic cardiomyopathy. There is strong evidence to support the role of ICDs for the primary prevention of sudden death in this population. However, in Canada and the United States, ICDs are underutilized.

Critical pathways are algorithms that improve health care delivery and clinical outcomes while reducing practice variability. The use of a critical pathway to assess a patient's eligibility for an ICD may increase the appropriate use of this evidence-based technology.

ELIGIBILITY:
Inclusion Criteria:

* acute ST segment elevation myocardial infarction (STEMI)
* candidate for percutaneous revascularization
* permanent residents of British Columbia, Canada

Exclusion Criteria:

* patients with heart disease or a comorbid illness who have a documented life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Referral for ICD Assessment | 1 year

SECONDARY OUTCOMES:
Rate of ICD Implantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: S Cowan, MD, MSc, Study Director — St. Paul's Hospital, Vancouver, British Columbia; A Ignaszewski, MD, Study Director — St. Paul's Hospital, Vancouver, British Columbia; C Kerr, MD, Principal Investigator — St. Paul's Hospital, Vancouver, British Columbia; S Tung, MD, Study Director — St. Paul's Hospital, Vancouver, British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada